CLINICAL TRIAL: NCT01069120
Title: A Phase III Multicenter Extension Study Evaluating the Safety of 25 and 50 mg Proellex® in the Treatment of Women Who Have Completed ZPU-301, ZPU-302, ZPU-303, or ZPU-304
Brief Title: Safety of 25 and 50 mg Proellex® in the Treatment of Women With Symptomatic Uterine Fibroids
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Repros stopped study due to safety and FDA placed study on hold
Sponsor: Repros Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZPU-307
Record Dates: First submitted 2010-02-10; First posted 2010-02-17 (Estimated); Results first posted 2014-08-21 (Estimated); Last update posted 2014-08-21 (Estimated); Status verified 2014-08

CONDITIONS: Uterine Fibroids
Keywords: Uterine Fibroids
MeSH Terms: conditions — Leiomyoma | interventions — telapristone acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 50 mg Proellex® (Active Comparator): 2, 25 mg capsules
  Interventions: Drug: Proellex
- 25 mg Proellex® (Active Comparator): 1, 25 mg capsule
  Interventions: Drug: Proellex

INTERVENTIONS:
Drug: Proellex — 2, 25 mg capsules once per day
  Other Names: CDB-4124
  Arms: 50 mg Proellex®
Drug: Proellex — 1, 25 mg capsule once per day
  Other Names: CDB-4124
  Arms: 25 mg Proellex®

SUMMARY:
Safety and efficacy study of 25 and 50 mg doses of Proellex

DETAILED DESCRIPTION:
The study is intended to provide more abundant safety and efficacy data of both the 25 and 50 mg doses of Proellex than ZPU-301, ZPU-302, ZPU-303 and ZPU-304 alone.

ELIGIBILITY:
Inclusion Criteria:

* At least 1 uterine fibroid must be identifiable and measurable by Transvaginal Ultrasound (TVU)
* Subject has a menstrual cycle lasting from 20 to 40 days.
* Subject must have satisfactorily completed all study visits from the previous study in which she participated: ZPU-301, ZPU-302, ZPU-303, or ZPU-304

Exclusion Criteria:

* Subjects who have not participated in 1 of the previous Repros studies: ZPU-301, ZPU-302, ZPU-303, or ZPU-304.
* Subjects who met treatment stopping rules as per the DILI Guidance requirements while participating in ZPU-301, ZPU-302, ZPU-303, or ZPU-304

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2009-04; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andre vanAS, PhD, Md, Study Director — Repros Therapeutics Inc.
Locations (4):
- United States (4):
  - Visions Clinical Research, Boynton Beach, Florida
  - Insignia Clinical Research (Tampa Bay Women's Center), Tampa, Florida
  - Advances in Health Inc, Houston, Texas
  - The Women's Hospital of Texas, Clinical Research Center, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Proellex®: 25 or 50 mg capsules once per day
Period: Overall Study
Arm/Group | Proellex®
Started | 27
Completed | 0
Not Completed | 27
Not completed — Study prematurely terminated | 27

BASELINE CHARACTERISTICS:
Population: Study prematurely terminated
Groups:
- Total: Total of all reporting groups
Arm/Group | 50 mg Proellex® | 25 mg Proellex® | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical [Count of Participants; unit: Participants]
Sex: Female, Male [Count of Participants; unit: Participants]
Region of Enrollment [Number; unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: To Assess the Incidence of Adverse Events (AE) and Serious Adverse Events (SAEs)
Time Frame: During two 4 month treatment periods
Arm/Group | 50 mg Proellex® | 25 mg Proellex®
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: No adverse events data is available.
Arm/Group | 50 mg Proellex® | 25 mg Proellex®
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The study was prematurely terminated for safety reasons (Proellex studies were put on clinical hold due to liver toxicity). Sponsor was unable to pay vendor, and was therefore not provided with any study data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to publication, Investigator shall submit to the Sponsor a copy of any proposed publication. Sponsor shall have sixty (60) days to review the proposed publication for possible disclosure of Sponsor's Confidential Information and, upon request of Sponsor, Investigator shall delete any of Sponsor's Confidential Information or withhold submission of such publication to allow Sponsor to protect its intellectual property rights